CLINICAL TRIAL: NCT04680767
Title: Disposition of [¹⁴C]-LY3502970 Following Oral Administration in Healthy Male Participants
Brief Title: A Study of LY3502970 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17784; J2A-MC-GZGF (Other: Eli Lilly and Company); 2020-003160-60 (EudraCT Number)
Record Dates: First submitted 2020-12-21; First posted 2020-12-23 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- [¹⁴C]-LY3502970 (Experimental): A single dose of LY3502970 and [¹⁴C]-LY3502970 administered orally.
  Interventions: Drug: LY3502970; Drug: [¹⁴C]-LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally.
Drug: [¹⁴C]-LY3502970 — Administered orally.

SUMMARY:
The main purpose of this study is to measure how much of the study drug gets into the bloodstream and how long it takes the body to eliminate it. This study will involve a single dose of ¹⁴C radiolabelled LY3502970. This means that a radioactive substance will be incorporated into the study drug. The purposes are to investigate the study drug and its breakdown products and to find out how much of these pass from blood into urine and feces. The study will last up to 8 weeks (maximum).

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males
* Body weight within 50 and 100 kilograms (kg), inclusive, and body mass index within the range 18.0 and 32.0 kilograms per square meter (kg/m²) (inclusive)

Exclusion Criteria:

* Females
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product (IP); or of interfering with the interpretation of data
* Have a history of Gilbert's syndrome or have total bilirubin level (TBL) above upper limit of normal (ULN) at screening
* Have evidence of significant active neuropsychiatric disease, as determined by the investigator
* Have had any exposure to LY3502970 or any other glucagon-like peptide-1 (GLP-1) analogs, or other related compounds within the prior 3 months, or any history of allergies to these medications
* Are currently enrolled in a clinical study involving an investigational product (IP) or any other type of medical research judged not to be scientifically or medically compatible with this study
* Have participated, within the last 3 months, in a clinical study involving an IP. If the previous IP has a long half-life, 5 half-lives or 3 months (whichever is longer) should have passed, prior to check-in
* Have participated in any clinical trial involving a radiolabeled IP within 12 months prior to check-in
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Have had exposure to significant diagnostic, therapeutic, or employment-related radiation within 12 months prior to dosing (e.g., serial x-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring)

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-07-03 (Actual); Study Completion 2021-07-03 (Actual)

PRIMARY OUTCOMES:
Fecal Excretion of LY3502970 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 17 after administration of study drug
  Fecal Excretion of LY3502970 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Urinary Excretion of LY3502970 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 17 after administration of study drug
  Urinary Excretion of LY3502970 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK): Area under the Concentration-Time Curve (AUC) of LY3502970 | Predose up to Day 17 after administration of study drug
  Plasma PK: AUC of LY3502970
Plasma PK: Maximum Concentration (Cmax) of LY3502970 | Predose up to Day 17 after administration of study drug
  Plasma PK: Cmax of LY3502970
Plasma and Whole Blood PK of Radioactivity: AUC | Predose up to Day 17 after administration of study drug
  Plasma and Whole Blood PK of Radioactivity: AUC
Plasma and Whole Blood PK of Radioactivity: Cmax | Predose up to Day 17 after administration of study drug
  Plasma and Whole Blood PK of Radioactivity: Cmax
Relative Abundance of LY3502970 and it's Metabolites in Plasma, Feces, and Urine | Predose up to Day 17 after administration of study drug
  Relative Abundance of LY3502970 and it's Metabolites in Plasma, Feces, and Urine

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No